CLINICAL TRIAL: NCT01484782
Title: Developing Accessible Telehealth Programs for Hypertensive Patients in Latin America
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, John Piette, Professor, University of Michigan, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UM-00047263
Record Dates: First submitted 2011-11-30; First posted 2011-12-02 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2015-04

CONDITIONS: Hypertension
Keywords: Hypertension; Telephone Care Management; Blood pressure; Medication adherence; Interactive Voice Response (IVR); Cloud computing
MeSH Terms: conditions — Hypertension; Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Interactive Voice Response (IVR) calls (Experimental): Weekly automated telephone assessment and behavior change calls focused on blood pressure management. The experimental group will receive a weekly 10-minute automated phone call to their telephone for disease assessment and self-care support for 6 weeks. In-home blood pressure cuffs were provided for measurement of blood pressure throughout the study.
  Interventions: Behavioral: Interactive Voice Response (IVR) automated calls
- Usual care (No Intervention): This group received results of blood pressure readings. PCP referrals. Educational materials about hypertension and self-management. At follow-up, patients received home blood pressure monitoring cuffs.

INTERVENTIONS:
Behavioral: Interactive Voice Response (IVR) automated calls — Interactive Voice Response (IVR) is a type of automated telephone call. Weekly automated telephone assessment and behavior change calls focused on blood pressure management will be sent to the experimental group. They will receive a weekly 10-minute automated phone call to their telephone for disease assessment and self-care support for 6 weeks. In-home blood pressure cuffs were provided for measurement of blood pressure throughout the study.
  Arms: Interactive Voice Response (IVR) calls

SUMMARY:
The purpose of this study is to evaluate the feasibility of utilizing an interactive voice response (IVR) system to supplement hypertension self-management for patients in underdeveloped regions in Mexico and Honduras. Weekly disease assessment calls included hypertension self-management suggestions and support to patients. The impact on patients' blood pressure levels and other secondary outcomes were evaluated.

DETAILED DESCRIPTION:
Background: Three quarters of all cardiovascular disease-related deaths occur in low- to middle- income countries. In addition, there are more than 1 billion people worldwide at risk of a serious cardiovascular event due to high blood pressure, high serum cholesterol levels and/or diabetes. In Latin America, hypertensive-related heart disease is among the top ten causes of death. Inadequacies in health care service access and treatment quality along with high rates of poverty, only work to exacerbate the problem.

Objectives/Aims: Based on prior study and other previous projects conducted in Santa Cruz de Yojoa, the purpose of the study is to evaluate the short-term feasibility and impact of an automated phone system in monitoring and improving hypertension among patients from semi-rural communities in Mexico and Honduras. The specific aims are: (1) to evaluate the feasibility (acceptability and usage rates) of a program including weekly disease assessment calls that include self-management suggestions and support among patients with hypertension; (2) to evaluate the program's impact on patients' blood pressure levels and other secondary outcomes; and (3) to discuss with local clinical, community, and health policy leaders the potential for expansion of this telemedicine program to other underdeveloped regions throughout the world and as well as its possible efficacy for other chronic diseases beyond cardiovascular diseases.

Methods: Adult hypertensive patients who receive care from participating clinics affiliated with Yojoa International Medical Center in Santa Cruz de Yojoa, Honduras and the Diabetes Center clinics in Pachuca and Real del Monte, Mexico, will be recruited for this study. 200 patients (100 from each clinic site), including adult men and women (up to 100 from each clinic) between the ages of 18 and 80 who have high blood pressure and who see their primary care doctor at one of the participating clinics will be screened and enrolled in this program. The patient may choose to enroll with a family member or friend (a "Care Partner") for disease management support throughout the study. Blood pressure will be taken by researchers at baseline, and at the six-week follow-up.

Participants will be randomized to receive written information about blood pressure control versus weekly automated telephone assessment and behavior change calls focused on blood pressure management. The intervention group will receive a weekly 10-minute automated phone call to their cell phone for disease assessment and self-care support for 6 weeks. Intervention patients also will be provided with in-home cuffs for measurement of blood pressure throughout the study. During patients' automated calls, they will be asked questions about their hypertension, medication, and self-care. Based on the patient's self-report, they will receive targeted suggestions for how to improve their hypertension self- care. The intervention patient's CarePartner (if applicable) will receive a weekly update via automated phone call or email, which will give that informal caregiver a summary of the enrolled patient's health and provide him/her with suggestions for addressing the needs of the patient and supporting the patient's self-care.

Urgent alerts for patients with critical health problems will be provided, via email, to the research team plus the clinic so that follow-up with a clinician can take place. The intervention will last six weeks, after which the patient will have a follow-up visit with the research team and will complete a survey about the program. The control group will be enrolled just as the intervention group; however, the control group will not receive automated phone calls or a blood pressure monitor over the six-week study period.

ELIGIBILITY:
Inclusion Criteria:

* Hypertension (for diabetic patients: systolic blood pressure 130 or greater; for non-diabetic patients: systolic blood pressure 140 or greater)
* Access to a functional telephone
* Able to respond to automated telephone calls

Exclusion Criteria:

* No access to a functional telephone
* Diagnosis of cancer with less than a six month life expectancy
* Severe mental illness as reported by their clinical team

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2011-05; Primary Completion 2011-11 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Systolic blood pressure | 6 weeks

SECONDARY OUTCOMES:
Self-reported health status | 6 weeks
Medication adherence | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: John D Piette, PhD, Principal Investigator — University of Michigan
Locations (2):
- Yojoa International Medical Center, Santa Cruz de Yojoa, Cortés Department, Honduras
- Remedi Diabetes Clinic, Pachuca, Hidalgo, Mexico